CLINICAL TRIAL: NCT06578897
Title: A Post-Market, Retrospective Study to Collect Clinical Outcomes From Patients Who Have Undergone Revision Total Knee Arthroplasty Using Medacta GMK Revision With 3D Metal Tibial and Femoral Cones.
Brief Title: A Post-Market, Retrospective Study on 3D Metal Tibial and Femoral Cones
Status: Completed | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: MUSA-CONES1-2023
Record Dates: First submitted 2024-08-21; First posted 2024-08-30 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: 3D Metal Tibial and Femoral cones — * To collect retrospective clinical outcomes and data on revision TKAs using Medacta GMK Revision with 3D metal tibial and femoral cones
  * Evaluate the patient reported functionality of the operated knee
  * Evaluate the clinical and radiological performance
  * Evaluate safety of the cones
  * Evaluate survivorship of revisions using tibial and femoral cones

SUMMARY:
GMK Revision Knee System is part of the Medacta GMK® (Global Medacta Knee) Total Knee System and is indicated when a higher level of varus/valgus constraint is needed. The external shape of the GMK® Revision femoral component is identical to that of GMK® Primary. The GMK® Revision differs from GMK® Primary by three important design features:

i. The addition of a box which allows a stem to be inserted into the femoral canal; ii. The addition of screw lugs so that augments can be placed on the distal and posterior resections, and; iii. The box which also allows various levels of constraint to be added to the polyethylene insert. The tibial component offers the ability to place augments.

Indications for Use:

The GMK® Total Knee System is designed for cemented use in total knee arthroplasty if there is evidence of sufficient sound bone to seat and support the components.

This knee replacement system is indicated in the following cases:

* Severely painful and/or disabled joint as a result of arthritis, traumatic arthritis, rheumatoid arthritis or polyarthritis
* Avascular necrosis of femoral condyle
* Post traumatic loss of joint configuration
* Primary implantation failure
* Ligamentous Instability

Tibial augments are to be attached to the tibial baseplate with both the fixing cylinders and bone cement. In case a semi-constrained liner is used, an extension stem must be implanted both on the tibial and on the femoral component.

GMK® Revision femoral components are manufactured of Cobalt Chromium Molybdenum (CoCrMo) according to ISO 5832-4:1996, Implants for Surgery- Metallic materials - Part 4: Cobalt-Chromium-Molybdenum Casting Alloy, the same as the GMK® Primary femoral components. They have an asymmetric patellar groove (left and right) with different radii of curvature in coronal plane as well as non-parallel anterior and posterior cuts (wedge shape). The GMK® Revision posterior stabilized femoral components are designed for use without cruciate ligaments when additional stability is required to prevent subluxation of the femur to the tibia in flexion, same as the GMK® Primary femoral components.

In case of severe bone loss, the tibial cones and femoral cones may be used to respectively reinforce the proximal tibia cavity and the distal femoral cavity, providing structural support and load redistribution on the remaining bone. Being an integral part of revision TKA for patients with such bone loss, the clinical outcomes for revision TKAs using the cone components are important for the knowledge regarding performance and survivorship of the Revision TKA as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Subjects underwent revision total knee replacement for any type of etiology (Osteoarthritis, Avascular necrosis, Rheumatoid Arthritis, Post-traumatic Arthritis, Polyarthritis, Primary implantation failure, Infection, Ligamentous Instability)
* Subjects must have received a Medacta GMK Revision component using 3D metal tibial and femoral cones
* Must be at minimum 1 year (12 months) post-treatment
* No age limit criteria

Exclusion Criteria:

* Subjects with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device
* Subjects that were incarcerated at the time of surgery.
* History of alcoholism
* On chemotherapy or radiation therapy during the time of interest
* Habitual use of narcotic pain medications prior to surgery or after surgery for reasons other than knee pain
* History of a metabolic disorder affecting the skeletal system other than osteoarthritis or osteoporosis
* History of chronic pain issues for reasons other than knee pain
* Progressive local or systemic infection during time of interest
* Muscular loss, neuromuscular disease, or vascular deficiency of the affected limb
* Obesity or excessive weight of subject

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The total expected number of subjects to be included in this study is a minimum number of 50. This number has been estimated according to the number of surgeries that have been performed and is considered in-line with observational studies published in literature.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
To collect retrospective clinical outcomes and data on revision TKAs using Medacta GMK Revision with 3D metal tibial and femoral cones | 1 year
  Oxford Knee Score (OKS) is a 12-item patient-reported PRO specifically designed and developed to assess function and pain after total knee replacement (TKR) surgery (arthroplasty).
  The overall score for the OKS is acquired by simply summing the scores received for individual questions. This results in a continuous score ranging from 0 (most severe symptoms/problems) to 48 (least severe).
To collect retrospective clinical outcomes and data on revision TKAs using Medacta GMK Revision with 3D metal tibial and femoral cones | 1 year
  Forgotten Joint Score (FJS) is a 12-question patient-reported outcomes measure created to measure a patient's awareness of their artificial joint.
  The FJS responses "never," "almost never," "seldom," "sometimes," and "mostly" translate into a 5-point Likert-response format translated linearly into a summative range from 0 to 100 scale with high values translating to the patient successfully "forgetting" about their joint during activities of daily living
To collect retrospective clinical outcomes and data on revision TKAs using Medacta GMK Revision with 3D metal tibial and femoral cones | 1 year
  Knee Injury and Osteoarthritis Outcome Score (KOOS) s a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury.
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures.

SECONDARY OUTCOMES:
Evaluate the clinical and radiological performance | 1 year
  standard x-ray exam performed preoperatively and postoperatively before discharge from hospital and during follow-up visits
Evaluate safety of the cones | through study completion, an average of 1 year
  Any complication occurred during the study
Evaluate survivorship of revisions using tibial and femoral cones | 1 year
  % survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No